CLINICAL TRIAL: NCT05734040
Title: Phase 2a, Randomized, Double-blind (Double-dummy), Double Placebo-controlled, Parallel-group Study to Evaluate the Immunogenicity and the Safety of the Concomitant Administration of OVX836 Influenza Vaccine and Quadrivalent Inactivated Influenza Vaccines (QIVs: Fluarix Tetra and Afluria Quad) Given Intramuscularly as 2 Separate Injections Into Opposite Arms, in Comparison to the Concomitant Administration of Quadrivalent Inactivated Influenza Vaccines and Placebo, and OVX836 and Placebo Given the Same Way in Healthy Subjects Aged 18 to 60 Years.
Brief Title: Immunogenicity and Safety of the Concomitant Administration of OVX836 Influenza Vaccine, Quadrivalent Inactivated Influenza Vaccines and Placebo in Healthy Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); Mater Misericordiae Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-006
Record Dates: First submitted 2023-02-09; First posted 2023-02-17 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized (1:1:1:1:1:1) into 6 groups of 100 subjects to receive:
  * First group: OVX836 480µg and Fluarix Tetra at commercial dose administered intramuscularly concomitantly into opposite arms.
  * Second group: OVX836 480µg and Afluria Quad at commercial dose administered intramuscularly concomitantly into opposite arms.
  * Third group: OVX836 480µg, concomitantly administered with placebo, intramuscularly into opposite arms.
  * Fourth group: Fluarix Tetra at commercial dose, concomitantly administered with placebo, intramuscularly into opposite arms.
  * Fifth group: Afluria Quad at commercial dose, concomitantly administered with placebo, intramuscularly into opposite arms.
  * Sixth group: placebo administered intramuscularly as two concomitant injections into opposite arms.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- OVX836 480µg + Fluarix Tetra at commercial dose (Experimental): OVX836: Adjuvant-free recombinant influenza candidate vaccine based on Nucleoprotein of the influenza virus. One single administration intramuscularly of 480µg dose on Day 1 AND Fluarix Tetra: Inactivated and purified split influenza vaccine. One single administration intramuscularly in the opposite arm on Day 1.
  Interventions: Biological: OVX836 480µg; Biological: Fluarix Tetra
- OVX836 480µg + Afluria Quad at commercial dose (Experimental): OVX836: Adjuvant-free recombinant influenza candidate vaccine based on Nucleoprotein of the influenza virus. One single administration intramuscularly of 480µg dose on Day 1 AND Afluria Quad: Inactivated and purified split influenza vaccine. One single administration intramuscularly in the opposite arm on Day 1.
  Interventions: Biological: OVX836 480µg; Biological: Afluria Quad
- Fluarix Tetra at commercial dose + Placebo (Active Comparator): Fluarix Tetra: Inactivated and purified split influenza vaccine. One single administration intramuscularly in the opposite arm on Day 1.
  AND Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50 milliliter. One single administration intramuscularly of a 0.8 milliliter dose in the opposite arm on Day 1.
  Interventions: Biological: Fluarix Tetra; Biological: Placebo
- Afluria Quad at commercial dose + Placebo (Active Comparator): Afluria Quad: Inactivated and purified split influenza vaccine. One single administration intramuscularly on Day 1.
  AND Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50 milliliter. One single administration intramuscularly of a 0.8 milliliter dose in the opposite arm on Day 1.
  Interventions: Biological: Afluria Quad; Biological: Placebo
- OVX836 480µg + Placebo (Placebo Comparator): OVX836: Adjuvant-free recombinant influenza candidate vaccine based on Nucleoprotein of the influenza virus. One single administration intramuscularly of 480µg dose on Day 1 AND Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50 milliliter. One single administration intramuscularly of a 0.8 milliliter dose in the opposite arm on Day 1.
  Interventions: Biological: OVX836 480µg; Biological: Placebo
- Placebo + Placebo (Placebo Comparator): Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50 milliliter. One single administration intramuscularly of a 0.8 milliliter dose on Day 1 AND Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50 milliliter. One single administration intramuscularly of a 0.8 milliliter dose in the opposite arm on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: OVX836 480µg — One single administration intramuscularly at Day 1
  Arms: OVX836 480µg + Afluria Quad at commercial dose; OVX836 480µg + Fluarix Tetra at commercial dose; OVX836 480µg + Placebo
Biological: Fluarix Tetra — One single administration intramuscularly at Day 1
  Arms: Fluarix Tetra at commercial dose + Placebo; OVX836 480µg + Fluarix Tetra at commercial dose
Biological: Afluria Quad — One single administration intramuscularly at Day 1
  Arms: Afluria Quad at commercial dose + Placebo; OVX836 480µg + Afluria Quad at commercial dose
Biological: Placebo — One single administration intramuscularly at Day 1
  Arms: Afluria Quad at commercial dose + Placebo; Fluarix Tetra at commercial dose + Placebo; OVX836 480µg + Placebo; Placebo + Placebo

SUMMARY:
The present study OVX836-006 aims principally to:

* Confirm feasibility of the concomitant administration of the vaccines under normal clinical conditions, i.e. as two separate concomitant injections into opposite arms;
* Introduce an additional representative brand of Quadrivalent Inactivated Influenza Vaccines ;
* Demonstrate the absence of interaction between OVX836 and Quadrivalent Inactivated Influenza Vaccines on the Hemagglutinin response;
* Demonstrate the absence of interaction between OVX836 and Quadrivalent Inactivated Influenza Vaccines on the nucleoprotein response;
* Evaluate the absolute vaccine efficacy of OVX836 compared to placebo in order to corroborate the efficacy signals previously detected in the OVX836 previous studies;
* Evaluate the combined vaccine efficacy of OVX836 + Quadrivalent Inactivated Influenza Vaccines versus OVX836 + placebo, and versus double placebo.

DETAILED DESCRIPTION:
Phase 2a, randomized, double-blind, double placebo-controlled, parallel-group study to evaluate the immunogenicity and the safety of the concomitant administration of :

* OVX836 influenza vaccine and Fluarix Tetra;
* OVX836 influenza vaccine and Afluria Quad;
* Fluarix Tetra and placebo;
* Afluria Quad and placebo;
* OVX836 influenza vaccine and placebo;
* Placebo and Placebo; given intramuscularly as 2 separate injections into opposite arms in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female subjects, as determined by medical history and medical examination.
3. Aged 18 to 60 years.
4. Subjects who have received at least two doses of a licensed severe acute respiratory syndrome Coronavirus 2 vaccine.
5. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures.
6. Able to read, understand and complete an electronic diary and electronic patient reported outcome, and availability of a person who can complete the electronic diary/electronic patient reported outcome in case of illness.

Exclusion Criteria:

1. Subjects with a body mass index ≤19 kg/m² or ≥40 kg/m² on the day of vaccination.
2. Previous influenza vaccination within 6 months before the day of vaccination or planned to receive influenza vaccination during the whole study period.
3. Any known or suspected immunodeficient conditions.
4. Past or current history of significant autoimmune diseases, as judged by the Investigator.
5. Known or suspected infection with human immunodeficiency virus, hepatitis C virus, or hepatitis B virus.
6. Current history of significant uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases, as judged by the Investigator.
7. Planned, recent (<6 months since completion) or ongoing gender reassignment during the study.
8. Female subjects: pregnant, breast-feeding or of childbearing potential without appropriate contraceptive methods in place for 2 months before enrolment, or with positive pregnancy test on the day of vaccination. Appropriate contraceptive methods are to be maintained until the end of the trial. Appropriate contraceptive methods are defined by the Clinical Trial Facilitation Group as follow: "Contraceptive methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include: combined (estrogen- and progestogencontaining) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable intrauterine device, intrauterine hormone-releasing system), bilateral tubal occlusion, vasectomized partner and/or sexual abstinence (refraining from heterosexual intercourse)."
9. Having received another vaccination within 3 months prior to the day of study vaccination for live attenuated vaccines, or within 1 month prior to the day of study vaccination for inactivated vaccines, except Coronavirus Disease 2019 vaccine.
10. Planning to receive other vaccines during the first 28 days following the study vaccine administration.
11. Having received a Coronavirus Disease 2019 vaccination within 2 weeks prior to the day of study vaccination.
12. Planning to receive Coronavirus Disease 2019 vaccine during the first week (within 7 days) following the study vaccine administration. An interval of preferably 14 days is recommended.
13. Administration of any investigational (including OVX836) or non-registered drug or vaccine within 3 months prior to the administration of study vaccines, or planned administration of any such product during the whole study period.
14. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination, or planned to receive such product during the whole study period.
15. Presence of an acute febrile illness on the day of planned vaccination (oral temperature >38.0°C; temporary exclusion criterion).
16. Long Coronavirus Disease, either ongoing or recently recovered.
17. Presence of a condition in the ear-nose-throat area, such as nasal septum deviation, atrophic rhinitis, etc., that could render nasal and nasopharyngeal swabs more difficult to perform, or increase the risk of bleeding; to be confirmed by medical history question and inspection of nasal passage.
18. Presence of tattoos at the level of one of the deltoid muscle.
19. Past or current history of any progressive or severe uncontrolled neurological disorder, seizure disorder or Guillain-Barré syndrome.
20. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
21. Past (stopped less than 6 months before enrolment) or current smoking habit above 10 cigarettes per day.
22. Past (stopped less than 6 months before enrolment) or current history of alcohol abuse or use of recreational drugs.
23. Treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800μg/day beclomethasone or equivalent; occasional inhaled corticosteroids for asthma therapy are allowed), radiation treatment, cytotoxic drugs, or current or recent (within 30 days before study entry) chronic or prolonged (>10 days) use of systemic non-steroidal anti-inflammatory drugs, acetylsalicylic acid, paracetamol, ibuprofen, interferon, immunomodulators, allergy shots, as judged by the Investigator. Occasional, non-continuous use of acetylsalicylic acid, paracetamol, ibuprofen or non-steroidal anti-inflammatory drugs on an as-needed basis is allowed.
24. Prophylactic or therapeutic use of any anti(retro)virals by systemic route during the study. Topical application is allowed.
25. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to kanamycin, eggs (especially ovalbumin and chicken proteins), neomycin, polymyxin, formaldehyde and octoxinol-9 (triton-X-100).
26. Any contraindication to intramuscular administration, as judged by the Investigator.
27. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study, or pose additional risk to the subjects due to participation in the study, either directly or through any treatments administered for that illness.
28. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse (or assimilated), parent, child or sibling, whether biological or legally adopted.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 478 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Number of seroconversion determined using Hemagglutination-Inhibition assay, for the four influenza strains contained in the Quadrivalent Inactivated Influenza Vaccines. | At Day 29 versus pre-injection baseline (Day 1)
  Seroconversion is defined as a negative pre-vaccination Hemagglutination-Inhibition assay titer and post-vaccination Hemagglutination-Inhibition assay titer ≥1:40, or a fourfold increase in Hemagglutination-Inhibition assay titer between pre- and post-vaccination timepoints.
Proportion of subjects achieving a titer ≥1:40 at Day 29 determined using Hemagglutination-Inhibition assay, for the four influenza strains contained in the Quadrivalent Inactivated Influenza Vaccine. | At Day 29
Number of Hemagglutination-Inhibition assay titers geometric mean ratios >2.5 for the four influenza strains contained in the Quadrivalent Inactivated Influenza Vaccines. | At Day 29 versus pre-injection baseline (Day 1)
Proportion of subjects reporting solicited local (Injection site redness, Injection site swelling, Injection site pain) and systemic signs and symptoms (Fatigue, Headache, Arthralgia, Malaise, Myalgia, Fever) | During 7 days after vaccine administration
Proportion of subjects reporting unsolicited Adverse Events | During 29 days after vaccine administration
Proportion of subjects reporting Serious Adverse Events | During the whole study duration, 180 days

SECONDARY OUTCOMES:
Hemagglutination-Inhibition assay geometric mean titers for each of the four strains contained in the Quadrivalent Inactivated Influenza Vaccines. | At Day 1 (pre-injection baseline) and Day 29
Number of laboratory-confirmed influenza A or B cases. | During the whole study duration, 180 days
Severity scores of Influenza-Like-Illness cases (as per Flu-PRO questionnaire) | During the whole study duration, 180 days
Cell-mediated immune response in terms of change of Nucleoprotein-specific T-cell frequencies in Peripheral Blood Mononuclear Cells, measured by Interferon Gamma Enzyme-Linked Immunospot Assay. | At Day 8 versus pre-injection baseline (Day 1)
Geometric Mean Titer of anti-Nucleoprotein immunoglobulin G (Enzyme-Linked Immunosorbent Assay, serum). | At Day 1, Day 8 and Day 29
Proportion of subjects with an increase (four-fold) in anti-Nucleoprotein Immunoglobulin G (Enzyme-Linked Immunosorbent Assay, serum) titer. | At Day 29 with respect to pre-injection baseline (Day 1)

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (9):
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Emeritus Research Sydney, Sydney, New South Wales
  - Paratus Clinical Research Western Sydney, Sydney, New South Wales
  - Paratus Clinical Research Brisbane, Brisbane, Queensland
  - Mater Misericordiae Limited, Brisbane, Queensland
  - UniSC Clinical Trials Moreton Bay, Morayfield, Queensland
  - University of Sunshine Coast, Sippy Downs, Queensland
  - CMAX Fusion Clinical Research, Adelaide, South Australia
  - Emeritus, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No